CLINICAL TRIAL: NCT05331729
Title: Evaluation of the Value of 18F-Fluoromisonidazole (18F-FMISO) Positron Emission Tomography Hypoxia Imaging in Idiopathic Pulmonary Fibrosis - a Non-randomized Proof-of-concept Study Comparing Patients with Idiopathic Pulmonary Fibrosis and Healthy Subjects
Brief Title: Evaluation of the Value of 18F-Fluoromisonidazole (18F-FMISO) Positron Emission Tomography Hypoxia Imaging in Idiopathic Pulmonary Fibrosis
Acronym: FIPOXY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: BELTRAMO_APJ_2019
Record Dates: First submitted 2022-04-04; First posted 2022-04-18 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with idiopathic pulmonary fibrosis (Experimental)
  Interventions: Radiation: FMISO-PET Protocol
- Healthy volunteers (Active Comparator)
  Interventions: Radiation: FMISO-PET Protocol

INTERVENTIONS:
Radiation: FMISO-PET Protocol — * injection of 18F-FMISO
  * Monitoring for 2 h
  * PET scan (30 min) 2h post injection
  * Monitoring for 2h
  * PET (30min) 4h post injection
  * Discharge of the subject with appropriate recommendations after a PET/CT

SUMMARY:
Idiopathic pulmonary fibrosis (IPF) is a rare, chronic, lethal disease of unknown etiology and with a variable course. There is currently no test in routine care that can assess both the anatomical and functional damage of the disease at an early stage. This is the first human study in IPF to evaluate the value of a non-invasive tracer, 18F-fluoromisonidazole (18F-FMISO), targeting hypoxia in IPF patients.

This is a Phase I, proof-of-concept, single-center, open-label, parallel group study.

It will include 2 groups:

* 1 group of 10 IPF patients
* 1 group of 10 healthy volunteers matched to IPF patients for age and gender

ELIGIBILITY:
Inclusion Criteria:

For all patients (IPF and healthy volunteers) :

* Person who has given written consent
* Age ≥ 50 years
* Absence of disease, comorbidity, or treatment that may interfere with the evaluation of the study objective, as decided by the investigator

For patients with IPF only:

* Diagnosis of IPF according to the criteria of the current international recommendations (ATS/ERS/JRS/ALAT of 2011) and validated in a multi-disciplinary meeting in a Competence or Reference Center
* Patients who have had a high-resolution thoracic CT scan less than 1 month previously as part of the management of their disease
* Patients who have had a PFT less than 1 month previously as part of the management of their disease

For healthy volunteers only:

* Absence of functional respiratory signs - absence of dyspnea on exertion and at rest and absence of chronic cough.
* Normal clinical examination with no crackles on pulmonary auscultation
* No personal history of chronic hypoxemic respiratory disease

Exclusion Criteria:

* Person who is not covered by national health insurance
* Cancer or history of cancer in the past 5 years (except basal cell skin cancer)
* Chronic lung disease other than IPF or a history incompatible with the diagnosis of idiopathic pulmonary fibrosis (thoracic radiotherapy, pneumotoxic chemotherapy, etc.)
* Exacerbation of IPF during treatment
* Active smoking
* Patient requiring long-term oxygen therapy (excluding ambulatory oxygen therapy alone)
* Contraindication to PET or CT scan or presence of a condition disturbing the interpretation :

  * known allergy to 18F-FMISO
  * pregnancy or breastfeeding
  * claustrophobia
  * uncontrolled type I/II diabetes (HbA1c >7%)
  * surgical intervention in the previous month
  * Radiotherapy session in the previous 3 months
  * concomitant granulomatous condition (sarcoidosis type) or pulmonary inflammation
* Moderate or severe renal insufficiency (GFR < 70 ml/min/1.73 m²)
* Person under legal protection (curatorship, guardianship)
* Adult unable to express consent
* SECONDARY EXCLUSION CRITERIA only for healthy volunteers

  * Abnormal 6 min walk test at screening
  * Abnormal PFT at screening with FVC ≤ 80% of predicted value and DLCO ≤ 75% of predicted value

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2025-02-20 (Actual); Study Completion 2025-02-20 (Actual)

PRIMARY OUTCOMES:
Lung SUVmean of 18F-FMISO measured in PET | At baseline
  Comparison in IPF patients and healthy volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No